CLINICAL TRIAL: NCT01154127
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Two-period Cross-over Study to Assess the Effect of 50µg Inhaled NVA237 on Exercise Endurance in Patients With Moderate to Severe COPD
Brief Title: Effect of NVA237 on Exercise Endurance in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: GLOW3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237A2310; 2010-018597-20 (EudraCT Number)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: NVA237; COPD; bronchodilator; exercise endurance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NVA237 followed by Placebo (Experimental): Period 1: 50 μg NVA237 via NEOHALER inhaler device for 21 days
  Period 2: Matching placebo via NEOHALER inhaler device for 21 days
  The washout period ran for 14 to 28 days between treatment periods. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study.
  Salbutamol (albuterol) was used as rescue medication throughout the study.
  Interventions: Drug: NVA237; Drug: Placebo
- Placebo followed by NVA237 (Experimental): Period 1: Matching placebo of NVA237 via NEOHALER inhaler device for 21 days
  Period 2: 50 μg NVA237 via NEOHALER inhaler device for 21 days
  The washout period ran for 14 to 28 days between treatment periods. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study.
  Salbutamol (albuterol) was used as rescue medication throughout the study.
  Interventions: Drug: NVA237; Drug: Placebo

INTERVENTIONS:
Drug: NVA237 — 50 μg via NEOHALER inhaler device single dose dry powder inhaler (SDDPI) once daily
Drug: Placebo — Matching placebo via NEOHALER inhaler device single dose dry powder inhaler (SDDPI) once daily

SUMMARY:
The ability for patients with COPD to exercise is limited due to the deterioration of their lung function. NVA237 is being developed to treat COPD. This study is designed to look at how well NVA237 improves the ability to exercise in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed an Informed Consent Form prior to initiation of any study-related procedure
* Patients with moderate to severe stable COPD (clinical diagnosis in compliance with GOLD 2008)
* Current or ex-smokers with a smoking history ≥ 10 pack years. (Ten pack-years were defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.).
* Patients with a post-bronchodilator FEV1 ≥ 40 and < 70% of the predicted normal, and postbronchodilator FEV1/FVC < 0.7 during screening. (Post referred to the highest post-bronchodilator value after inhalation of 80 μg ipratropium bromide)
* Increase in FEV1 from pre- to post-bronchodilator assessment of ≥ 5%

Exclusion Criteria:

* Pregnant women or nursing mothers
* Women of child-bearing potential
* Patients who had a COPD exacerbation (whether hospitalized or not) in the 6 weeks prior to Visit 1 or between Visit 1 and Visit 4
* Patients who had a lower respiratory tract infection in the 6 weeks prior to Visit 1
* Patients requiring long term oxygen therapy on a daily basis for chronic hypoxemia
* Patients with resting (5 min) oxygen SaO2 (or SpO2) saturation on room air of < 85%
* Patients with a maximum workload (Wmax) value < 20 W (as determined by the incremental cycle endurance test) at Visit 2.
* Patients whose exercise endurance time at sub-maximal workload was above 25 min at baseline
* Patients with a clinically significant abnormality on the screening or baseline ECG who in the judgment of the investigator would have been at potential risk if enrolled into the study
* Patients with a history of long QT syndrome or whose QTc was prolonged (> 450 ms for males and > 470 ms females) at screening (Fredericia's correction)

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Spartanburg Medical Research, 485 Simuel Road, Spartanburg, South Carolina, United States
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Woehrendamm
- Novartis Investigative Site, Verona, Italy
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Manchester, United Kingdom

REFERENCES:
- [Derived] Beeh KM, Singh D, Di Scala L, Drollmann A. Once-daily NVA237 improves exercise tolerance from the first dose in patients with COPD: the GLOW3 trial. Int J Chron Obstruct Pulmon Dis. 2012;7:503-13. doi: 10.2147/COPD.S32451. Epub 2012 Jul 31. PMID 22973092

RESULTS

PARTICIPANT FLOW:
Groups:
- NVA237 Followed by Placebo: Period 1: 50 μg NVA237 via NEOHALER inhaler device for 21 days.
  Period 2: Matching placebo via NEOHALER inhaler device for 21 days
  The washout period ran for 14 to 28 days between treatment periods. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study.
  Salbutamol (albuterol) was used as rescue medication throughout the study.
- Placebo Followed by NVA237: Period 1: Matching placebo of NVA237 via NEOHALER inhaler device for 21 days
  Period 2: 50 μg NVA237 via NEOHALER inhaler device for 21 days.
  The washout period ran for 14 to 28 days between treatment periods. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study.
  Salbutamol (albuterol) was used as rescue medication throughout the study.
Period: Period 1 (21 Days)
Arm/Group | NVA237 Followed by Placebo | Placebo Followed by NVA237
Started | 55 | 53
Completed | 52 | 47
Not Completed | 3 | 6
Not completed — Adverse Event | 3 | 4
Not completed — Withdrawal by Subject | 0 | 2
Period: Washout (14 - 28 Days)
Arm/Group | NVA237 Followed by Placebo | Placebo Followed by NVA237
Started | 52 | 47
Completed | 49 | 47
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Abnormal Test Procedure | 1 | 0
Period: Period 2 (21 Days)
Arm/Group | NVA237 Followed by Placebo | Placebo Followed by NVA237
Started | 49 | 47
Completed | 49 | 46
Not Completed | 0 | 1
Not completed — Protocol Deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 Followed by Placebo | Placebo Followed by NVA237 | Total
Number analyzed (Participants) | 55 | 53 | 108
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.50) | 59.7 (8.78) | 60.5 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Exercise Endurance Time During a Sub-maximal Constant-load Cycle Ergometry Test (SMETT) After 3 Weeks (Day 21) of Treatment
Description: SMETT is an exercise procedure where the patient cycles at 80% of the maximum workload (Wmax )value achieved at the Incremental exercise test. During this test, the patient will cycle at a constant load. Exercise endurance time was from commencement of loaded pedaling to stopping exercise. The analysis-of covariance model included the sequence, period, and treatment as fixed factors, the baseline value as covariate and the patient as a random effect.
Time Frame: Day 21
Population: Pharmacodynamics (PD) set consisted of participants who completed at least one treatment period, had an evaluable PD assessment on Day 21 of this period and had no major protocol deviation impacting the primary PD assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Groups:
- NVA237: Participants received NVA237 50 μg once daily delivered via the NEOHALER inhaler device device for 3 weeks (21 days).
  The washout period ran for 14 to 28 days between treatment periods. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study.
  Salbutamol (albuterol) was used as rescue medication throughout the study.
- Placebo: Participants received Placebo 50 μg once daily delivered via the NEOHALER inhaler device device for 3 weeks (21 days).
  The washout period ran for 14 to 28 days between treatment periods. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study.
  Salbutamol (albuterol) was used as rescue medication throughout the study.
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 96 | 96
seconds | 505.63 [466.59 to 544.68] | 416.70 [377.76 to 455.64]

2. Secondary Outcome: Isotime Inspiratory Capacity (IC) During Sub-maximal Constant-load Cycle Ergometry Test (SMETT) After 3 Weeks of Treatment
Description: Isotime is the last matching timepoint in the submaximal exercise tolerance test (SMETT) at which for both periods the patient has a test result. The analysis-of covariance model included the sequence, period, and treatment as fixed factors, the baseline value as covariate and the patient as a random effect.
Time Frame: Day 21
Population: Pharmacodynamics (PD) set consisted of participants who completed at least one treatment period, had an evaluable PD assessment on Day 21 of this period and had no major protocol deviation impacting primary the PD assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 92 | 92
Liters | 2.22 [2.15 to 2.31] | 2.02 [1.95 to 2.08]

3. Secondary Outcome: Inspiratory Capacity (IC) at Rest (1 Hour Post Dose) and at Peak (End of Exercise) During Sub-maximal Constant-load Cycle Ergometry Test (SMETT) After 3 Weeks of Treatment
Description: IC at peak was observed using spirometry. However, two different methodologies (whole body plethysmography (Bodybox) and spirometry) were used to observe IC at rest.
  The analysis of covariance model included the sequence, period, and treatment as fixed factors, the baseline value as covariate and the patient as a random effect.
Time Frame: Day 21
Population: Pharmacodynamics (PD) set consisted of participants who completed at least one treatment period, had an evaluable PD assessment on Day 21 of this period and had no major protocol deviation impacting the primary PD assessment. "n" indicates number of participants with observation at each time-point.
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 99 | 96
Litres
  IC at peak (Spirometry), Day 21 (n = 93, 90) | 2.22 [2.16 to 2.28] | 2.03 [1.97 to 2.10]
  IC at rest (Bodybox) Day 21 (n= 97, 96) | 2.49 [2.40 to 2.59] | 2.26 [2.17 to 2.35]
  IC at rest (Spirometry), Day 21 (n= 98, 96) | 2.39 [2.33 to 2.45] | 2.17 [2.10 to 2.23]

4. Secondary Outcome: Peak and Trough (24 h Post Dose) Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC)
Description: FEV1 is the amount of air that can be exhaled in one second. FEV1 was measured with spirometry conducted according to internationally accepted standards.
  FVC is the volume of air that can forcibly be blown out after full inspiration and is used in spirometry tests.
  The trough effects of Day 1 treatment are derived from values prior to morning dosing on the next treatment day (Day 2 of the corresponding period).
  The analysis-of covariance model included the sequence, period, and treatment as fixed factors, the baseline value as covariate and the patient as a random effect.
Time Frame: Day 21
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 99 | 96
Litres
  FEV1 at peak, Day 21 | 1.60 [1.56 to 1.64] | 1.35 [1.31 to 1.39]
  FEV1 at trough, Day 21 | 1.44 [1.40 to 1.48] | 1.33 [1.29 to 1.37]
  FVC at peak, Day 21 | 3.37 [3.30 to 3.44] | 3.00 [2.93 to 3.06]
  FVC at trough, Day 21 | 3.17 [3.11 to 3.23] | 2.96 [2.90 to 3.02]

5. Secondary Outcome: Slow Vital Capacity (SVC) and Total Lung Capacity (TLC)
Description: Vital Capacity is the amount of air that can be forcibly exhaled from the lungs after a full inhalation. Slow Vital Capacity (SVC) test is performed by having the patient slowly and completely blow out all of the air from their lungs.
  Total Lung Capacity (TLC) is the best vital capacity plus residual volume. Whole body plethysmography (Bodybox) was used to measure SVC and TLC. The trough effects of Day 1 treatment are derived from values prior to morning dosing on the next treatment day (Day 2 of the corresponding period).
Time Frame: Day 21
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 99 | 96
Litres
  SVC at trough, Day 21 (n= 98, 96) | 3.21 [3.14 to 3.27] | 3.14 [3.07 to 3.21]
  SVC at peak, Day 21 (n= 97, 96) | 3.40 [3.33 to 3.47] | 3.14 [3.07 to 3.21]
  TLC at trough, Day 21 (n= 98, 96) | 6.99 [6.88 to 7.09] | 7.17 [7.07 to 7.28]
  TLC at peak, Day 21 (n= 97, 96) | 6.86 [6.75 to 6.97] | 7.10 [6.99 to 7.21]

6. Secondary Outcome: Specific Airways Conductance (SGaw)
Description: SGaw is a measure of how hard it is to get air into the lungs, measured by (Sec(-1)*kP). Whole body plethysmography (Bodybox) was used to measure SGaw.
  The analysis-of covariance model included the sequence, period, and treatment as fixed factors, the baseline value as covariate and the patient as a random effect.
Time Frame: Day 21
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: litres/(Second*kpa); kpa = kilopascal
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 99 | 96
litres/(Second*kpa); kpa = kilopascal
  SGaw at trough, Day 21 (n= 98, 96) | 0.48 [0.45 to 0.51] | 0.40 [0.38 to 0.43]
  SGaw at peak, Day 21 (n= 97, 96) | 0.66 [0.63 to 0.70] | 0.42 [0.39 to 0.46]

7. Secondary Outcome: Exertional Dyspnea (Borg CR10 Scale) During Sub-maximal Constant-load Cycle Ergometry Test (SMETT) After 3 Weeks Treatment
Description: The Borg CR10 Scale consists of 12-point score that the patients pointed to so as to indicate their level of dyspnea before and during exercise testing (where 0 indicates no breathlessness at all and 12 indicates maximum breathlessness).
  A reduction in this score indicates an improvement. The analysis-of covariance model included the sequence, period, and treatment as fixed factors, the baseline value as covariate and the patient as a random effect.
Time Frame: Day 21
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 93 | 93
units on a scale | 5.64 [5.05 to 6.23] | 6.80 [6.20 to 7.39]

8. Secondary Outcome: Leg Discomfort (Borg CR10 Scale) During Sub-maximal Constant-load Cycle Ergometry Test (SMETT) After 3 Weeks Treatment
Description: The modified Borg CR10 Scale consists of 12-point score that the patients pointed to so as to indicate their level of leg discomfort before and during exercise testing (where 0 indicates no breathlessness at all and 12 indicates maximum breathlessness).
  A reduction in this score indicates an improvement. The analysis-of covariance model included the sequence, period, and treatment as fixed factors, the baseline value as covariate and the patient as a random effect.
Time Frame: Day 21
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 93 | 93
units on a scale | 6.21 [5.67 to 6.76] | 7.05 [6.51 to 7.60]

9. Secondary Outcome: Exercise Endurance Time During a Sub-maximal Constant-load Cycle Ergometry Test (SMETT) on Treatment Day 1
Description: as for outcome 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 96 | 94
Seconds | 490.92 [458.45 to 523.38] | 447.78 [415.09 to 480.48]

ADVERSE EVENTS:
Description: All patients as randomized who received at least one dose of study drug are included in the safety analysis set.
Groups:
- NVA237; Placebo: Period 1: 50 μg NVA237 via NEOHALER inhaler device for 21 days
  Period 2: Matching placebo via NEOHALER inhaler device for 21 days
  The washout period ran for 14 to 28 days between treatment periods. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study.
  Salbutamol (albuterol) was used as rescue medication throughout the study.
Arm/Group | NVA237 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/102 | 0/102
Other Adverse Events (participants affected / at risk) | 0/102 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=102) | Placebo (N=102)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.